CLINICAL TRIAL: NCT02073149
Title: Comparison of Home Fortification With Two Iron Formulations in Kenyan Children Protected Against Malaria by Artemisinin-based Combination Therapy: a Placebo-controlled Non-inferiority Trial
Brief Title: Safe and Efficacious Iron for Children in Kenya
Acronym: SEICK
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Maseno University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSHTM-2542
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2014-02

CONDITIONS: Anaemia
Keywords: Iron; Anemia; Sodium Fe(III)-ethylenediaminetetraacetic acid (NaFeEDTA); Ferrous compounds; Child, preschool; Kenya
MeSH Terms: conditions — Anemia | interventions — Iron; Fe(III)-EDTA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low-dose iron as NaFeEDTA (Active Comparator): Daily point-of-care fortification of (complementary) foods with 3 mg iron as NaFeEDTA.
  Interventions: Dietary Supplement: Low-dose iron as NaFeEDTA
- Conventional dose iron as ferrous salt (Active Comparator): Daily point-of-care fortification of (complementary) foods with 12.5 mg iron as encapsulated ferrous fumarate.
  Interventions: Dietary Supplement: Conventional dose iron as ferrous salt
- Placebo (Placebo Comparator): Daily point-of-care fortification of (complementary) foods with placebo.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Low-dose iron as NaFeEDTA — Daily home fortification for 30 days with 3 mg iron as NaFeEDTA, vitamin A (300 RE μg as retinyl palmitate) and 5 mg zinc (as gluconate)
  Arms: Low-dose iron as NaFeEDTA
Dietary Supplement: Conventional dose iron as ferrous salt — Daily home fortification for 30 days with 12.5 mg iron as encapsulated ferrous fumarate, vitamin A (300 RE μg as retinyl palmitate) and 5 mg zinc (as gluconate)
  Arms: Conventional dose iron as ferrous salt
Dietary Supplement: Placebo — Daily home fortification for 30 days with vitamin A (300 RE μg as retinyl palmitate) and 5 mg zinc (as gluconate)
  Arms: Placebo

SUMMARY:
This study will determine whether the haemoglobin response to daily home fortification for 30 days with 3mg iron as NaFeEDTA is non-inferior to 12.5 mg iron as encapsulated ferrous fumarate.

DETAILED DESCRIPTION:
Background: Fortification of local complementary foods and supplementation with micronutrient powders including iron has been shown to prevent anaemia. Iron can cause complaints (diarrhoea, constipation, etc.) related to oxidative stress in the intestine, however, and at doses conventionally used for daily supplementation, iron can increase rates of malaria and diarrhoea. A lower dose of iron (3mg/day) as NaFEEDTA can reduce these adverse effects whilst having similar or superior efficacy in improving iron status as conventional-dose iron (12.5mg) as ferrous salts.

Objective: The primary aim is to compare daily home fortification with 3mg iron as NaFeEDTA versus 12.5 mg iron as encapsulated ferrous fumarate regarding haemoglobin concentration at the end of the 30-day fortification period.

Methods: Rural children aged 12-36 months (n=324) will receive albendazole and praziquantel against helminth infections, and preventive chemotherapy against malaria with dihydroartemisinin-piperaquine. They will subsequently be randomised to daily home fortification for 30 days with sachets containing either a) 3 mg iron as NaFeEDTA; b) 12.5 mg iron as encapsulated ferrous fumarate; or c) placebo. Parents or guardians will be instructed to mix the contents of the sachets with solid or semi-solid, ready-prepared foods. Adherence will be assessed by an electronic monitoring and time-recording device in the cap of a dispensing bottle containing the sachets. At the end of the 30-day fortification period, a venous blood sample will be collected to measure indicators of iron status and inflammation. Children who received iron will continue to be followed for a maximum of 120 days after randomisation to estimate the time point when ≥10% of children has developed severe anaemia (haemoglobin concentration <70 g/L).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 12-36 months;
2. Residing in the study area;
3. Planning to be in the area for the duration of the intervention and follow-up;
4. Study protocol accepted and informed consent given by at least one parent or guardian

Exclusion Criteria:

1. Known or reported allergy to dihydroartemisinin, piperaquine, benzimidazole drugs or praziquantel;
2. A sibling from the same household already randomised to intervention;
3. Severely malnourished (weight-for-height z-score < -3 SD) (for ethical reasons);
4. Presence of fever (axillary temperature ≥ 37.5 ºC) (to avoid inflammation-induced effects on iron status markers);
5. Presence of reported or suspected systemic disorder (e.g. HIV infection, sickle cell disease) (to avoid inflammation-induced effects on iron status markers and to avoid attrition);
6. Missed one or several doses of the 3-day course of dihydroartemisinin-piperaquine (to ensure that participants are protected against malaria for the duration of the iron intervention);
7. No blood sample collected, or blood volume collected < 5 mL;
8. Haemoglobin concentration < 70 g/L (to prevent severe anaemia).

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 338 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin concentration | End of the 30-day fortification period

SECONDARY OUTCOMES:
Iron status | End of the 30-day fortification period
  Iron status will be assessed by plasma concentrations of ferritin and soluble transferrin receptor
Serum concentration of non-transferrin bound iron | 3 hours after ingesting the first fortificant dose
Faecal calprotectin concentration | End of the 30-day fortification period
  Faecal calprotectin concentration is used as an indicator of intestinal inflammation
P. falciparum infection | End of the 30-day fortification period
  P. falciparum infection will be defined as the presence of either asexual parasites in blood smears or parasite antigens (either histidine-rich protein-2, or Plasmodium lactate dehydrogenase) in whole blood
Adherence to intervention | End of the 30-day fortification period
  Adherence will be defined for each individual as the number of days that the dispensing bottle has been opened during the 30-day intervention period

OTHER OUTCOMES:
Haemoglobin concentration | Single measurement between 30 and 100 days after randomisation
  At various time points in the post-intervention period, we will sample children without replacement to measure their haemoglobin concentration. Taking into account our wish to restrict phlebotomies during the post-intervention period to a single occasion per child, we will withdraw the child from further study. These measurements should allow us to estimate the time point when ≥10% of children has developed severe anaemia (haemoglobin concentration <70 g/L).

CONTACTS AND LOCATIONS:
Overall Officials: Hans Verhoef, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Maseno University, Maseno, Nyanza Province, Kenya

REFERENCES:
- [Derived] Teshome EM, Oriaro VS, Andango PEA, Prentice AM, Verhoef H. Adherence to home fortification with micronutrient powders in Kenyan pre-school children: self-reporting and sachet counts compared to an electronic monitoring device. BMC Public Health. 2018 Feb 1;18(1):205. doi: 10.1186/s12889-018-5097-2. PMID 29391008
- [Derived] Teshome EM, Prentice AM, Demir AY, Andang'o PEA, Verhoef H. Diagnostic utility of zinc protoporphyrin to detect iron deficiency in Kenyan preschool children: a community-based survey. BMC Hematol. 2017 Jul 27;17:11. doi: 10.1186/s12878-017-0082-z. eCollection 2017. PMID 28770094
- [Derived] Teshome EM, Andang'o PEA, Osoti V, Terwel SR, Otieno W, Demir AY, Prentice AM, Verhoef H. Daily home fortification with iron as ferrous fumarate versus NaFeEDTA: a randomised, placebo-controlled, non-inferiority trial in Kenyan children. BMC Med. 2017 Apr 28;15(1):89. doi: 10.1186/s12916-017-0839-z. PMID 28449690